CLINICAL TRIAL: NCT05489237
Title: A First-in-human (FIH) Study of IDRX-42 in Participants With Metastatic and/or Unresectable Gastrointestinal Stromal Tumors (GIST) [Study ID: StrateGIST 1]
Brief Title: First-in-human Study of IDRX-42 in Participants With Metastatic and/or Unresectable Gastrointestinal Stromal Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: IDRx Inc. - A GSK Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 300382; IDRX-42-001 (Other: IDRx Inc. - A GSK Company); 2024-514930-19-00 (EU CTIS Number)
Record Dates: First submitted 2022-07-28; First posted 2022-08-05 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Gastrointestinal Neoplasms; Gastrointestinal Stromal Tumor (GIST); Digestive System Disease; Gastrointestinal Diseases; Metastatic Cancer
Keywords: GIST; IDRX; IDRX-42; Strate; StrateGIST; StrateGIST 1
MeSH Terms: conditions — Gastrointestinal Neoplasms; Gastrointestinal Stromal Tumors; Digestive System Diseases; Gastrointestinal Diseases; Neoplasm Metastasis | interventions — IDRX-42

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Escalation (Phase I) (Experimental): Participants should have advanced (metastatic and/or surgically unresectable) GIST, following failure of at least prior imatinib therapy due to progression of GIST.
  Interventions: Drug: IDRX-42
- (Phase 1b) Cohort 1 - Participants with GIST progression after first-line imatinib therapy (Experimental): Participants with advanced GIST who have had GIST progression after first-line imatinib only (second line therapy setting) and refused or are ineligible for other standard of care (SOC) therapies.
  Interventions: Drug: IDRX-42
- (Phase 1b): Cohort 2 - Participants with GIST progression after 2 or more lines of TKI therapy (Experimental): Participants with metastatic and/or surgically unresectable GIST following progression EITHER after sequential imatinib then sunitinib (third-line therapy setting) OR after imatinib, sunitinib, and then an additional TKI agent (i.e., regorafenib or ripretinib) (fourth-line therapy setting) OR after imatinib, sunitinib, regorafenib, and ripretinib (5th line or greater therapy).
  Interventions: Drug: IDRX-42
- (Phase 1b): Cohort 3 - Participants with GIST who are treatment naïve (Experimental): Participants with metastatic and/or surgically unresectable GIST who are treatment naïve (first line therapy) and refused or are ineligible for other standard of care (SOC) therapies.
  Interventions: Drug: IDRX-42
- (Phase 1b): Cohort 4 (Experimental): Participants with GIST progression who meet the same criteria as Cohort 2 (third line or greater TKI therapy) and have had prior treatment with investigational agents NB003 or THE-630 or a line of therapy of bezuclastinib plus sunitinib combination.
  Interventions: Drug: IDRX-42

INTERVENTIONS:
Drug: IDRX-42 — Administered at assigned doses and schedules once or twice daily in continuous cycles of 28 days each.

SUMMARY:
This is the first clinical trial of IDRX-42. The study is designed to evaluate the safety, tolerability, PK, and preliminary antitumor activity of IDRX-42 in adult participants with advanced (metastatic and/or surgically unresectable) GIST.

DETAILED DESCRIPTION:
This is a Phase 1/1b open-label, first-in-human FIH study of IDRX-42, an orally administered small molecule tyrosine kinase inhibitor. Eligible participants will have metastatic and/or surgically unresectable GIST. The study consists of 2 parts. Phase 1 comprises dose escalation to assess clinical and pharmacologic profile and safety/tolerability after failure of at least prior imatinib and support choice of the recommended phase 1b dose(s) and schedule(s) (RP1bDs)). Phase 1b expansion will enroll separate cohorts of participants defined by numbers of lines of prior GIST therapy at the selected RP1bD(s) to assess the preliminary antitumor effect of IDRX-42 and further characterize the safety profile of IDRX-42 at the RP1bD(s). In addition, a Concentration-QTc (C-QTc) substudy will be conducted in a subset of participants enrolled at selected sites in the study to characterize the effects of IDRX-42 on QTc and other ECG parameters in GIST patients.

ELIGIBILITY:
Inclusion Criteria:

Phase 1

1. Male or female participants ≥18 years of age
2. Histologically or cytologically confirmed metastatic and/or surgically unresectable GIST
3. Documented progression on imatinib (Phase 1)
4. Documented pathogenic mutation in KIT OR any PDGFRA mutation other than exon 18 mutations, determined through local testing
5. At least one measurable lesion by mRECIST v1.1 for participants with GIST
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Resolution of any toxicities from prior treatment(s) to ≤ Grade 1 by NCI CTCAE v5.0 criteria, or have resolved to baseline, at the time of first dose of study drug.
8. Willing and able to comply with scheduled visits, drug administration plan, laboratory tests, or other study procedures and study restrictions.

Additional for Phase 1b Exploratory Cohorts

1. For Cohort 1, progressed on imatinib only (second line therapy) and refused or are ineligible for other standard of care (SOC) therapies.
2. For Cohort 2, progressed on both imatinib and sunitinib (third line therapy) or progressed on imatinib, sunitinib, and an additional agent (i.e., regorafenib or ripretinib) (fourth line therapy) or progressed on imatinib, sunitinib, regorafenib, and ripretininb (fifth line or greater therapy)
3. For Cohort 3, treatment naïve (first line therapy) and refused or are ineligible for other standard of care (SOC) therapies.
4. For Cohort 4, met the same criteria as Cohort 2 (third line or greater) and have also had prior treatment with investigational agents NB003 or THE-630 or a line of therapy of bezuclastinib plus sunitinib combination.

Exclusion Criteria:

1. Any prior exposure to the following investigational agents NB003 or THE-630 or bezuclastinib plus sunitinib combination (except for participants treated in Cohort 4 of Phase 1b).
2. GIST with no documented mutation in both KIT and PDGFRA genes.
3. Primary brain malignancy or known untreated or active central nervous system metastases.
4. Has an active uncontrolled infection, including, but not limited to, the requirement for intravenous antibiotics.
5. Has significant, uncontrolled, or active cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2027-11-03 (Estimated); Study Completion 2027-11-03 (Estimated)

PRIMARY OUTCOMES:
Phase 1 (Dose Escalation) - Safety and Tolerability (Nature, incidence, and severity of any DLTs) | When participant completes 1 cycle (28 days) treatment with safety and tolerability assessment by investigators
Phase 1 (Dose Escalation) - Safety and Tolerability (Nature, incidence, and severity of any DLTs) | Approximately 18 months from first participant enrolled
Phase 1 (Dose Escalation) - Determination of the MTD and/or RP1bD(s) of orally administered IDRX-42 | Approximately 18 months from first participant enrolled
Phase 1 (Dose Escalation) - C-QTc sub-study: QTcF - concentration response analysis | At the end of Cycle 1 Day 1 and at the end of Cycle 2 Day 1 (each cycle is 28 days)
Phase 1b-Number of participants with TEAEs and with laboratory test results | Approximately 18 months
Phase 1b - Objective Response Rate (ORR) mRESIST v1.1 | Approximately 18 months
Phase 1b - C-QTcF sub-study: QTcF - concentration response analysis | At the end of Cycle 1 Day 1 and at the end of Cycle 2 Day 1 (each cycle is 28 days)

SECONDARY OUTCOMES:
Phase 1 (Dose Escalation)- Number of participants with non-DLT TEAEs and with laboratory test results | 6 months
Phase 1 (Dose Escalation) - ORR per mRECIST v1.1 | 6 months
Phase 1 (Dose Escalation) - Cmax; Maximum Observed Concentration of IDRX-42 | At the end of Cycle 1 Day 1 and at the end of Cycle 2 Day 1 (each cycle is 28 days)
Phase 1 (Dose Escalation) - Tmax; Time of First Occurrence of Maximum Plasma Concentration (Cmax) of IDRX-42 | At the end of Cycle 1 Day 1 and at the end of Cycle 2 Day 1 (each cycle is 28 days)
Phase 1 (Dose Escalation) - AUC 0-24; Area Under the Concentration-time Curve from Time Zero to 24 hours for IDRX-42 | At the end of Cycle 1 Day 1 and at the end of Cycle 2 Day 1 (each cycle is 28 days)
Phase 1 (Dose Escalation) - Duration of response (DOR) per mRECIST v1.1 | 6 months
Phase 1 (Dose Escalation) - Time to response (TTR) per mRECIST v1.1 | 6 months
Phase 1 (Dose Escalation) - Progression-free survival (PFS), per mRECIST v1.1 | 6 months
Phase 1 (Dose Escalation) - C-QTcF sub-study: QTcF, heart rate, PR, QRS interval at baseline, post baseline and change from baseline. | At the end of Cycle 1 Day 1 and at the end of Cycle 2 Day 1 (each cycle is 28 days)
Phase 1b- Duration of response (DOR) per mRECIST v1.1 | 18 months
Phase 1b - PFS per mRECIST v1.1 | 18 months
Phase 1b - Clinical benefit rate (CBR) per mRECIST v1.1 | 18 months
Phase 1b - TTR per mRECIST v1.1 | 18 months
Phase 1b - Cmax; Maximum Observed Concentration of IDRX-42 | At the end of Cycle 1 Day 1 and at the end of Cycle 2 Day 1 (each cycle is 28 days)
Phase 1b - Tmax; Time of First Occurrence of Maximum Plasma Concentration (Cmax) of IDRX-42 | At the end of Cycle 1 Day 1 and at the end of Cycle 2 Day 1 (each cycle is 28 days)
Phase 1b - AUC 0-24; Area Under the Concentration-time Curve from Time Zero to 24 hours for IDRX-42 | At the end of Cycle 1 Day 1 and at the end of Cycle 2 Day 1 (each cycle is 28 days)
Phase 1b - Overall survival | 18 months
Phase 1b C-QTc sub-study: QTcF, heart rate, PR, QRS interval at baseline, post baseline and change from baseline. | At the end of Cycle 1 Day 1 and at the end of Cycle 2 Day 1 (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (7):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Houston, Texas
- GSK Investigational Site, Leuven, Belgium
- China (3):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Wuhan
- France (4):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Villejuif
- Germany (2):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Essen
- GSK Investigational Site, Milan, Italy
- Japan (2):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Tokyo
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Rotterdam
- South Korea (2):
  - GSK Investigational Site, Seongnam-si Gyeonggi-do
  - GSK Investigational Site, Seoul
- GSK Investigational Site, Barcelona, Spain
- United Kingdom (2):
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, London